CLINICAL TRIAL: NCT04309240
Title: The Efficacy and Safety of Rivaroxaban for Thromboprophylaxis in High-risk Cancer Patients With Totally Implantable Access Ports: a Prospective Randomized Controlled Trial
Brief Title: Rivaroxaban for Thromboprophylaxis in High-risk Cancer Patients With Totally Implantable Access Ports
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: LiuZhou People's Hospital (Other)
Responsible Party: Principal Investigator, tingliu, Principal Investigator, LiuZhou People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY-1-2020-07-01
Record Dates: First submitted 2020-03-08; First posted 2020-03-16 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Rivaroxaban; Thromboprophylaxis; Cancer
Keywords: Prophylactic Anticoagulation; rivaroxaban; venous thrombosis; Totally Implantable Access Ports; cancer
MeSH Terms: conditions — Neoplasms; Venous Thrombosis | interventions — Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rivaroxaban (Experimental): oral Rivaroxaban 10mg per day for 90days
  Interventions: Drug: Rivaroxaban
- blank control (No Intervention): mechanical prophylaxis

INTERVENTIONS:
Drug: Rivaroxaban — Rivaroxaban 10mg orally per day for 90days
  Arms: rivaroxaban

SUMMARY:
Rivaroxaban has been developed in the various clinical settings.Although cancer-associated DVT or PE was included in previously programs, limited patients of the total populations were cancer patients with totally implantable access ports in these studies. In this sense, investigators feel that new oral anticoagulants should be re-investigated in this highly specific patients group.Therefore, investigators are planning to conduct a prospective study to estimate the efficacy and safety of rivaroxaban for thromboprophylaxis in high-risk cancer patients with totally implantable access ports.

ELIGIBILITY:
Eligibility Criteria:

1. Age 18-75 years;
2. Patients with malignant tumors who received implantable access ports for treatment;
3. Eastern Cooperative Oncology Group (ECOG) class 0-1;
4. will have a life expectancy > 3 months;
5. Expected survival of more than 6 months;
6. Khorana score ≥2 point.

Exclusion Criteria:

1. Patients with a history of allergies to rivaroxaban;
2. History of recent major or clinically relevant bleeding within the previous 4 weeks.
3. Patients with bleeding risks: thrombocytopenia (platelet count < 50*109/L), clinically significant active bleeding, active gastric ulcer disease, severe arterial hypertension, history of previous stroke; Inadequate renal function; creatinine clearance < 30 ml/min；
4. Inadequate hepatic function: aminotransferase > 3 times the upper limit of normal (ULN) (if liver metastasis, alanine aminotransferase > 5 times the ULN
5. Patients requiring strong cytochrome P450 3A4 (CYP3A4) inducers (rifampin, phenobarbital) or strong CYP3A4 inhibitors (HIV protease inhibitor, systemic ketoconazole) treatments.
6. Plan of treatment with bevacizumab or other anti-cancer drugs known to increase the bleeding risk.
7. Patients who have had anticoagulant drugs for any other reason.
8. Women who are pregnant or breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2020-03-08 (Estimated); Primary Completion 2022-03-08 (Estimated); Study Completion 2022-03-08 (Estimated)

PRIMARY OUTCOMES:
occurrence of venous thrombosis | From date of randomization until the date of occurrence of thrombosis or date of death from any cause, whichever came first, assessed up to 6 months
  detect the occurrence of venous thrombosis with ultrasound, venography if necessary.
occurrence of a major bleeding event. | From date of randomization until the date of occurrence of a major bleeding event or date of death from any cause, whichever came first, assessed up to 6 months
  define occurrence of major-bleeding event with ISTH standard
occurrence of clinically relevant non-major-bleeding, minor-bleeding or non-bleeding event | From date of randomization until the date of occurrence of events or date of death from any cause, whichever came first, assessed up to 6 months
  define occurrence of non-major-bleeding or minor-bleeding event with ISTH standard, evaluate the relevant adverse drug reaction with NCI CTCAE 5.0

CONTACTS AND LOCATIONS:
Overall Officials: yu bin, PHD, Study Chair — LiuZhou People's Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khorana AA, Soff GA, Kakkar AK, Vadhan-Raj S, Riess H, Wun T, Streiff MB, Garcia DA, Liebman HA, Belani CP, O'Reilly EM, Patel JN, Yimer HA, Wildgoose P, Burton P, Vijapurkar U, Kaul S, Eikelboom J, McBane R, Bauer KA, Kuderer NM, Lyman GH; CASSINI Investigators. Rivaroxaban for Thromboprophylaxis in High-Risk Ambulatory Patients with Cancer. N Engl J Med. 2019 Feb 21;380(8):720-728. doi: 10.1056/NEJMoa1814630. PMID 30786186
- [Background] Wang TF, Zwicker JI, Ay C, Pabinger I, Falanga A, Antic D, Noble S, Khorana AA, Carrier M, Meyer G. The use of direct oral anticoagulants for primary thromboprophylaxis in ambulatory cancer patients: Guidance from the SSC of the ISTH. J Thromb Haemost. 2019 Oct;17(10):1772-1778. doi: 10.1111/jth.14564. Epub 2019 Jul 28. No abstract available. PMID 31353841